CLINICAL TRIAL: NCT01039766
Title: The Efficacy of the Proximate Administration of Oxytocin After a Traumatic Event in Preventing the Development of Post Traumatic Stress Disorder
Brief Title: The Efficacy of a Single Dose of Intranasal Oxytocin in the Prevention of Post Traumatic Stress Disorder (PTSD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SHEBA-09-7128-AJW-CTIL
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: post traumatic stress disorder; prevention; oxytocin
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxytocin (Experimental)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo - saline nasal spray

INTERVENTIONS:
Drug: Oxytocin — A single intranasal administration of 40 IU of oxytocin will be given to patients up to 6 hours after a traumatic event, with consecutive follow up for 13 months.
  Other Names: syntocinon nasal spray
  Arms: oxytocin
Drug: placebo - saline nasal spray — A single intranasal administration of saline will be given to patients up to 6 hours after a traumatic event, with consecutive follow up for 13 months as the control to the oxytocin arm
  Other Names: saline nasal spray prepared by the hospital's pharmacy
  Arms: Placebo

SUMMARY:
This study is designed to test the hypothesis that a single administration of intranasal oxytocin within 6 hours post-trauma facilitates the physiological recovery for the trauma, thereby preventing the development of Post Traumatic Stress Disorder (PTSD) in the months following the event. In the absence of such treatment (i.e., under placebo conditions), we hypothesize that a greater proportion of persons will develop PTSD (i.e., fail to recover from acute effects).

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled trial in which trauma victims are randomized to receive a single intranasal administration of either Oxytocin (40IU) or placebo within the first six hours following trauma exposure. To provide a pre-treatment baseline, participants will receive a medical and psychological evaluation prior to treatment. After two weeks the research assistant or study psychiatrist will perform behavioral ratings and complete history details pertaining to PTSD risk factors. Participants will be assessed again by the study psychiatrist or research assistants at 1, 3, 6 and 13 months. Eligible subjects will include men and women over the age of 18, who have been exposed to an event meeting the DSM-IV "A.1" criterion for trauma exposure, and who provide written, informed consent to participate in the study. In order to recruit persons who are more likely to be at risk for the development of PTSD, we will only randomize persons expressing marked anxiety, emotional distress or dissociation, as assessed by the Visual Analog Scales. Potential participants will be recruited from trauma victims arriving at the Chaim Sheba Medical Center Emergency Room.

ELIGIBILITY:
Inclusion Criteria:

1. Persons over the age of 18, who have been exposed to an event meeting the DSM-IV "A.1" criterion for trauma exposure, expressing marked anxiety, and/ or emotional distress and/or dissociation, as assessed by the Visual Analog Scales
2. The traumatic event occured up to six hour prior to the arrival to the emergency room
3. The person can and is willing to provide written, informed consent to participate in the study.

Exclusion Criteria:

1. Physical injury that would contraindicate participation or interfere with a subject's ability to give informed consent or cooperate with the screening or collection of initial measures. Examples include severe burn injury, life-threatening medical or surgical condition, condition requiring surgical intervention under general anesthesia, as indicated by Abbreviated Injury Scale (AIS), or by clinical judgment;
2. Head injury involving confusion, loss of consciousness, or amnesia;
3. Medical conditions in which oxytocin administration might cause harm to the patient such as patients with a cardiovascular disease or intracranial mass.
4. Weight below 45 or above 100 kg.
5. Pregnancy (in suggestive cases, a pregnancy test will be performed);
6. Traumatic exposure that reflects ongoing victimization (e.g., domestic violence) to which the subject is likely to be re-exposed during the study period.
7. Overt psychopathology, intoxication, or under the influence of substances.
8. Evidence or history of schizophrenia, bipolar, other psychotic condition, autism;
9. Prior history of PTSD;
10. Current or past history of dementia, amnesia, or other cognitive disorder predating trauma exposure;
11. Assessed serious suicide risk.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-01 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is DSM-IV diagnosis of PTSD at the end of the trial. | 13 months

SECONDARY OUTCOMES:
The secondary outcome measure is the severity of PTSD as expressed by the Clinician Administered PTSD Scale (CAPS), at the end of the trial. | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Alzbeta Juven Wetzler, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Andrews B, Brewin CR, Rose S, Kirk M. Predicting PTSD symptoms in victims of violent crime: the role of shame, anger, and childhood abuse. J Abnorm Psychol. 2000 Feb;109(1):69-73. doi: 10.1037//0021-843x.109.1.69. PMID 10740937
- [Background] Beckner VE, Tucker DM, Delville Y, Mohr DC. Stress facilitates consolidation of verbal memory for a film but does not affect retrieval. Behav Neurosci. 2006 Jun;120(3):518-27. doi: 10.1037/0735-7044.120.3.518. PMID 16768603
- [Background] Davidson JR, Tupler LA, Wilson WH, Connor KM. A family study of chronic post-traumatic stress disorder following rape trauma. J Psychiatr Res. 1998 Sep-Oct;32(5):301-9. doi: 10.1016/S0022-3956(98)00016-8. PMID 9789209
- [Background] Koenen KC, Harley R, Lyons MJ, Wolfe J, Simpson JC, Goldberg J, Eisen SA, Tsuang M. A twin registry study of familial and individual risk factors for trauma exposure and posttraumatic stress disorder. J Nerv Ment Dis. 2002 Apr;190(4):209-18. doi: 10.1097/00005053-200204000-00001. PMID 11960081
- [Background] Kuhlmann S, Wolf OT. Arousal and cortisol interact in modulating memory consolidation in healthy young men. Behav Neurosci. 2006 Feb;120(1):217-23. doi: 10.1037/0735-7044.120.1.217. PMID 16492134
- [Background] Lupien SJ, Maheu F, Tu M, Fiocco A, Schramek TE. The effects of stress and stress hormones on human cognition: Implications for the field of brain and cognition. Brain Cogn. 2007 Dec;65(3):209-37. doi: 10.1016/j.bandc.2007.02.007. Epub 2007 Apr 26. PMID 17466428
- [Background] Stein MB, Jang KL, Taylor S, Vernon PA, Livesley WJ. Genetic and environmental influences on trauma exposure and posttraumatic stress disorder symptoms: a twin study. Am J Psychiatry. 2002 Oct;159(10):1675-81. doi: 10.1176/appi.ajp.159.10.1675. PMID 12359672
- [Background] Yehuda R, Bierer LM, Schmeidler J, Aferiat DH, Breslau I, Dolan S. Low cortisol and risk for PTSD in adult offspring of holocaust survivors. Am J Psychiatry. 2000 Aug;157(8):1252-9. doi: 10.1176/appi.ajp.157.8.1252. PMID 10910787
- [Background] Yehuda R, Halligan SL, Bierer LM. Relationship of parental trauma exposure and PTSD to PTSD, depressive and anxiety disorders in offspring. J Psychiatr Res. 2001 Sep-Oct;35(5):261-70. doi: 10.1016/s0022-3956(01)00032-2. PMID 11591428
- [Background] Yehuda R, Halligan SL, Grossman R. Childhood trauma and risk for PTSD: relationship to intergenerational effects of trauma, parental PTSD, and cortisol excretion. Dev Psychopathol. 2001 Summer;13(3):733-53. doi: 10.1017/s0954579401003170. PMID 11523857
- [Background] Yehuda R, Harvey PD, Buchsbaum M, Tischler L, Schmeidler J. Enhanced effects of cortisol administration on episodic and working memory in aging veterans with PTSD. Neuropsychopharmacology. 2007 Dec;32(12):2581-91. doi: 10.1038/sj.npp.1301380. Epub 2007 Mar 28. PMID 17392739
- [Background] Yehuda R. Post-traumatic stress disorder. N Engl J Med. 2002 Jan 10;346(2):108-14. doi: 10.1056/NEJMra012941. No abstract available. PMID 11784878
- [Background] Anisman H, Griffiths J, Matheson K, Ravindran AV, Merali Z. Posttraumatic stress symptoms and salivary cortisol levels. Am J Psychiatry. 2001 Sep;158(9):1509-11. doi: 10.1176/appi.ajp.158.9.1509. PMID 11532740
- [Background] Delahanty DL, Raimonde AJ, Spoonster E. Initial posttraumatic urinary cortisol levels predict subsequent PTSD symptoms in motor vehicle accident victims. Biol Psychiatry. 2000 Nov 1;48(9):940-7. doi: 10.1016/s0006-3223(00)00896-9. PMID 11074232
- [Background] Delahanty DL, Raimonde AJ, Spoonster E, Cullado M. Injury severity, prior trauma history, urinary cortisol levels, and acute PTSD in motor vehicle accident victims. J Anxiety Disord. 2003;17(2):149-64. doi: 10.1016/s0887-6185(02)00185-8. PMID 12614659
- [Background] Resnick HS, Yehuda R, Pitman RK, Foy DW. Effect of previous trauma on acute plasma cortisol level following rape. Am J Psychiatry. 1995 Nov;152(11):1675-7. doi: 10.1176/ajp.152.11.1675. PMID 7485635
- [Background] Yehuda R, Bryant R, Marmar C, Zohar J. Pathological responses to terrorism. Neuropsychopharmacology. 2005 Oct;30(10):1793-805. doi: 10.1038/sj.npp.1300816. PMID 16012535
- [Background] Yehuda R, McFarlane AC, Shalev AY. Predicting the development of posttraumatic stress disorder from the acute response to a traumatic event. Biol Psychiatry. 1998 Dec 15;44(12):1305-13. doi: 10.1016/s0006-3223(98)00276-5. PMID 9861473
- [Background] Yehuda R, LeDoux J. Response variation following trauma: a translational neuroscience approach to understanding PTSD. Neuron. 2007 Oct 4;56(1):19-32. doi: 10.1016/j.neuron.2007.09.006. PMID 17920012
- [Background] Charney DS, Deutch AY, Krystal JH, Southwick SM, Davis M. Psychobiologic mechanisms of posttraumatic stress disorder. Arch Gen Psychiatry. 1993 Apr;50(4):295-305. doi: 10.1001/archpsyc.1993.01820160064008. No abstract available. PMID 8466391
- [Background] Yehuda R, Halligan SL, Bierer LM. Cortisol levels in adult offspring of Holocaust survivors: relation to PTSD symptom severity in the parent and child. Psychoneuroendocrinology. 2002 Jan-Feb;27(1-2):171-80. doi: 10.1016/s0306-4530(01)00043-9. PMID 11750777
- [Background] Marmar CR, McCaslin SE, Metzler TJ, Best S, Weiss DS, Fagan J, Liberman A, Pole N, Otte C, Yehuda R, Mohr D, Neylan T. Predictors of posttraumatic stress in police and other first responders. Ann N Y Acad Sci. 2006 Jul;1071:1-18. doi: 10.1196/annals.1364.001. PMID 16891557
- [Background] Neylan TC, Brunet A, Pole N, Best SR, Metzler TJ, Yehuda R, Marmar CR. PTSD symptoms predict waking salivary cortisol levels in police officers. Psychoneuroendocrinology. 2005 May;30(4):373-81. doi: 10.1016/j.psyneuen.2004.10.005. Epub 2005 Jan 11. PMID 15694117
- [Background] Pariante CM, Nemeroff CB, Miller AH. Glucocorticoid receptors in depression. Isr J Med Sci. 1995 Dec;31(12):705-12. PMID 8543464
- [Background] Sautter FJ, Bissette G, Wiley J, Manguno-Mire G, Schoenbachler B, Myers L, Johnson JE, Cerbone A, Malaspina D. Corticotropin-releasing factor in posttraumatic stress disorder (PTSD) with secondary psychotic symptoms, nonpsychotic PTSD, and healthy control subjects. Biol Psychiatry. 2003 Dec 15;54(12):1382-8. doi: 10.1016/s0006-3223(03)00571-7. PMID 14675802
- [Background] Yehuda R, Engel SM, Brand SR, Seckl J, Marcus SM, Berkowitz GS. Transgenerational effects of posttraumatic stress disorder in babies of mothers exposed to the World Trade Center attacks during pregnancy. J Clin Endocrinol Metab. 2005 Jul;90(7):4115-8. doi: 10.1210/jc.2005-0550. Epub 2005 May 3. PMID 15870120
- [Background] Yehuda R, Teicher MH, Seckl JR, Grossman RA, Morris A, Bierer LM. Parental posttraumatic stress disorder as a vulnerability factor for low cortisol trait in offspring of holocaust survivors. Arch Gen Psychiatry. 2007 Sep;64(9):1040-8. doi: 10.1001/archpsyc.64.9.1040. PMID 17768269
- [Background] Cohen H, Zohar J, Gidron Y, Matar MA, Belkind D, Loewenthal U, Kozlovsky N, Kaplan Z. Blunted HPA axis response to stress influences susceptibility to posttraumatic stress response in rats. Biol Psychiatry. 2006 Jun 15;59(12):1208-18. doi: 10.1016/j.biopsych.2005.12.003. Epub 2006 Feb 3. PMID 16458266
- [Background] Harvey BH, Brand L, Jeeva Z, Stein DJ. Cortical/hippocampal monoamines, HPA-axis changes and aversive behavior following stress and restress in an animal model of post-traumatic stress disorder. Physiol Behav. 2006 May 30;87(5):881-90. doi: 10.1016/j.physbeh.2006.01.033. Epub 2006 Mar 6. PMID 16546226
- [Background] Kohda K, Harada K, Kato K, Hoshino A, Motohashi J, Yamaji T, Morinobu S, Matsuoka N, Kato N. Glucocorticoid receptor activation is involved in producing abnormal phenotypes of single-prolonged stress rats: a putative post-traumatic stress disorder model. Neuroscience. 2007 Aug 10;148(1):22-33. doi: 10.1016/j.neuroscience.2007.05.041. Epub 2007 Jul 17. PMID 17644267
- [Background] Mason JW, Giller EL, Kosten TR, Ostroff RB, Podd L. Urinary free-cortisol levels in posttraumatic stress disorder patients. J Nerv Ment Dis. 1986 Mar;174(3):145-9. doi: 10.1097/00005053-198603000-00003. PMID 3950596
- [Background] Yehuda R, Teicher MH, Trestman RL, Levengood RA, Siever LJ. Cortisol regulation in posttraumatic stress disorder and major depression: a chronobiological analysis. Biol Psychiatry. 1996 Jul 15;40(2):79-88. doi: 10.1016/0006-3223(95)00451-3. PMID 8793040
- [Background] Oquendo MA, Echavarria G, Galfalvy HC, Grunebaum MF, Burke A, Barrera A, Cooper TB, Malone KM, John Mann J. Lower cortisol levels in depressed patients with comorbid post-traumatic stress disorder. Neuropsychopharmacology. 2003 Mar;28(3):591-8. doi: 10.1038/sj.npp.1300050. Epub 2002 Aug 19. PMID 12629542
- [Background] Rohleder N, Joksimovic L, Wolf JM, Kirschbaum C. Hypocortisolism and increased glucocorticoid sensitivity of pro-Inflammatory cytokine production in Bosnian war refugees with posttraumatic stress disorder. Biol Psychiatry. 2004 Apr 1;55(7):745-51. doi: 10.1016/j.biopsych.2003.11.018. PMID 15039004
- [Background] Yehuda R. Current status of cortisol findings in post-traumatic stress disorder. Psychiatr Clin North Am. 2002 Jun;25(2):341-68, vii. doi: 10.1016/s0193-953x(02)00002-3. PMID 12136504
- [Background] Bremner JD, Southwick SM, Johnson DR, Yehuda R, Charney DS. Childhood physical abuse and combat-related posttraumatic stress disorder in Vietnam veterans. Am J Psychiatry. 1993 Feb;150(2):235-9. doi: 10.1176/ajp.150.2.235. PMID 8422073
- [Background] Marazziti D, Catena Dell'osso M. The role of oxytocin in neuropsychiatric disorders. Curr Med Chem. 2008;15(7):698-704. doi: 10.2174/092986708783885291. PMID 18336283
- [Background] Heinrichs M, Domes G. Neuropeptides and social behaviour: effects of oxytocin and vasopressin in humans. Prog Brain Res. 2008;170:337-50. doi: 10.1016/S0079-6123(08)00428-7. PMID 18655894
- [Background] Bartz JA, Hollander E. The neuroscience of affiliation: forging links between basic and clinical research on neuropeptides and social behavior. Horm Behav. 2006 Nov;50(4):518-28. doi: 10.1016/j.yhbeh.2006.06.018. Epub 2006 Aug 1. PMID 16884725
- [Background] Neumann ID. Involvement of the brain oxytocin system in stress coping: interactions with the hypothalamo-pituitary-adrenal axis. Prog Brain Res. 2002;139:147-62. doi: 10.1016/s0079-6123(02)39014-9. PMID 12436933
- [Background] Carter CS, Altemus M. Integrative functions of lactational hormones in social behavior and stress management. Ann N Y Acad Sci. 1997 Jan 15;807:164-74. doi: 10.1111/j.1749-6632.1997.tb51918.x. PMID 9071349
- [Background] Lightman SL, Young WS 3rd. Lactation inhibits stress-mediated secretion of corticosterone and oxytocin and hypothalamic accumulation of corticotropin-releasing factor and enkephalin messenger ribonucleic acids. Endocrinology. 1989 May;124(5):2358-64. doi: 10.1210/endo-124-5-2358. PMID 2785027
- [Background] Neumann ID, Johnstone HA, Hatzinger M, Liebsch G, Shipston M, Russell JA, Landgraf R, Douglas AJ. Attenuated neuroendocrine responses to emotional and physical stressors in pregnant rats involve adenohypophysial changes. J Physiol. 1998 Apr 1;508 ( Pt 1)(Pt 1):289-300. doi: 10.1111/j.1469-7793.1998.289br.x. PMID 9490853
- [Background] Stern JM, Goldman L, Levine S. Pituitary-adrenal responsiveness during lactation in rats. Neuroendocrinology. 1973;12(3):179-91. doi: 10.1159/000122167. No abstract available. PMID 4353345
- [Background] Thoman EB, Conner RL, Levine S. Lactation suppresses adrenal corticosteroid activity and aggressiveness in rats. J Comp Physiol Psychol. 1970 Mar;70(3):364-9. doi: 10.1037/h0028710. No abstract available. PMID 5461489
- [Background] Walker CD, Lightman SL, Steele MK, Dallman MF. Suckling is a persistent stimulus to the adrenocortical system of the rat. Endocrinology. 1992 Jan;130(1):115-25. doi: 10.1210/endo.130.1.1309321.
- [Background] Windle RJ, Wood S, Shanks N, Perks P, Conde GL, da Costa AP, Ingram CD, Lightman SL. Endocrine and behavioural responses to noise stress: comparison of virgin and lactating female rats during non-disrupted maternal activity. J Neuroendocrinol. 1997 Jun;9(6):407-14. doi: 10.1046/j.1365-2826.1997.00587.x. PMID 9229351
- [Background] Uvnas-Moberg K. Oxytocin may mediate the benefits of positive social interaction and emotions. Psychoneuroendocrinology. 1998 Nov;23(8):819-35. doi: 10.1016/s0306-4530(98)00056-0. PMID 9924739
- [Background] Uvnas-Moberg K, Ahlenius S, Hillegaart V, Alster P. High doses of oxytocin cause sedation and low doses cause an anxiolytic-like effect in male rats. Pharmacol Biochem Behav. 1994 Sep;49(1):101-6. doi: 10.1016/0091-3057(94)90462-6. PMID 7816858
- [Background] Lundeberg T, Uvnas-Moberg K, Agren G, Bruzelius G. Anti-nociceptive effects of oxytocin in rats and mice. Neurosci Lett. 1994 Mar 28;170(1):153-7. doi: 10.1016/0304-3940(94)90262-3. PMID 8041495
- [Background] Heinrichs M, Meinlschmidt G, Neumann I, Wagner S, Kirschbaum C, Ehlert U, Hellhammer DH. Effects of suckling on hypothalamic-pituitary-adrenal axis responses to psychosocial stress in postpartum lactating women. J Clin Endocrinol Metab. 2001 Oct;86(10):4798-804. doi: 10.1210/jcem.86.10.7919. PMID 11600543
- [Background] Uvnas-Moberg K. Neuroendocrinology of the mother-child interaction. Trends Endocrinol Metab. 1996 May-Jun;7(4):126-31. doi: 10.1016/1043-2760(96)00036-7. PMID 18406738
- [Background] Legros JJ, Chiodera P, Geenen V, Smitz S, von Frenckell R. Dose-response relationship between plasma oxytocin and cortisol and adrenocorticotropin concentrations during oxytocin infusion in normal men. J Clin Endocrinol Metab. 1984 Jan;58(1):105-9. doi: 10.1210/jcem-58-1-105. PMID 6315753
- [Background] Legros JJ, Chiodera P, Demey-Ponsart E. Inhibitory influence of exogenous oxytocin on adrenocorticotropin secretion in normal human subjects. J Clin Endocrinol Metab. 1982 Dec;55(6):1035-9. doi: 10.1210/jcem-55-6-1035. PMID 6290521
- [Background] Chiodera P, Coiro V. Oxytocin reduces metyrapone-induced ACTH secretion in human subjects. Brain Res. 1987 Sep 8;420(1):178-81. doi: 10.1016/0006-8993(87)90257-5. PMID 2823973
- [Background] Suh BY, Liu JH, Rasmussen DD, Gibbs DM, Steinberg J, Yen SS. Role of oxytocin in the modulation of ACTH release in women. Neuroendocrinology. 1986;44(3):309-13. doi: 10.1159/000124661. PMID 3027599
- [Background] House JS, Landis KR, Umberson D. Social relationships and health. Science. 1988 Jul 29;241(4865):540-5. doi: 10.1126/science.3399889.
- [Background] DeVries AC, Glasper ER, Detillion CE. Social modulation of stress responses. Physiol Behav. 2003 Aug;79(3):399-407. doi: 10.1016/s0031-9384(03)00152-5. PMID 12954434
- [Background] Henry JP, Wang S. Effects of early stress on adult affiliative behavior. Psychoneuroendocrinology. 1998 Nov;23(8):863-75. doi: 10.1016/s0306-4530(98)00058-4. PMID 9924741
- [Background] Insel TR, Young LJ. The neurobiology of attachment. Nat Rev Neurosci. 2001 Feb;2(2):129-36. doi: 10.1038/35053579. PMID 11252992
- [Background] Heinrichs M, Baumgartner T, Kirschbaum C, Ehlert U. Social support and oxytocin interact to suppress cortisol and subjective responses to psychosocial stress. Biol Psychiatry. 2003 Dec 15;54(12):1389-98. doi: 10.1016/s0006-3223(03)00465-7. PMID 14675803
- [Background] Winslow JT, Noble PL, Lyons CK, Sterk SM, Insel TR. Rearing effects on cerebrospinal fluid oxytocin concentration and social buffering in rhesus monkeys. Neuropsychopharmacology. 2003 May;28(5):910-8. doi: 10.1038/sj.npp.1300128. Epub 2003 Mar 26. PMID 12700704
- [Background] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222
- [Background] Kirsch P, Esslinger C, Chen Q, Mier D, Lis S, Siddhanti S, Gruppe H, Mattay VS, Gallhofer B, Meyer-Lindenberg A. Oxytocin modulates neural circuitry for social cognition and fear in humans. J Neurosci. 2005 Dec 7;25(49):11489-93. doi: 10.1523/JNEUROSCI.3984-05.2005. PMID 16339042
- [Background] Breslau N, Chilcoat HD, Kessler RC, Davis GC. Previous exposure to trauma and PTSD effects of subsequent trauma: results from the Detroit Area Survey of Trauma. Am J Psychiatry. 1999 Jun;156(6):902-7. doi: 10.1176/ajp.156.6.902. PMID 10360130
- [Background] Keane TM, Gerardi RJ, Lyons JA, Wolfe J. The interrelationship of substance abuse and posttraumatic stress disorder. Epidemiological and clinical considerations. Recent Dev Alcohol. 1988;6:27-48. doi: 10.1007/978-1-4615-7718-8_2. PMID 3283857
- [Background] Schumm JA, Briggs-Phillips M, Hobfoll SE. Cumulative interpersonal traumas and social support as risk and resiliency factors in predicting PTSD and depression among inner-city women. J Trauma Stress. 2006 Dec;19(6):825-36. doi: 10.1002/jts.20159. PMID 17195981
- [Background] Yehuda R. Biological factors associated with susceptibility to posttraumatic stress disorder. Can J Psychiatry. 1999 Feb;44(1):34-9. doi: 10.1177/070674379904400104. PMID 10076739
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873